CLINICAL TRIAL: NCT02177903
Title: Randomized, Prospective Study to Determine the Effects of Pre-warming on OR Patient Temperatures and Perioperative Surgical Outcomes
Brief Title: Study to Determine the Effects of Pre-warming on OR Patient Temperatures and Surgical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-05-013093
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Hypothermia
Keywords: hypothermia; surgical site infection; opioid usage; blood loss; pain severity; anxiety; Length of Stay
MeSH Terms: conditions — Hypothermia; Surgical Wound Infection; Hemorrhage; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bair PawsPatient Adjustable Warming System (Other): Bair PawsPatient Adjustable Warming System for active pre-warming
  Interventions: Device: Bair Paws Patient Adjustable Warming System
- Passive pre-warming (Other): Passive pre-warming
  Interventions: Device: Bair Paws Patient Adjustable Warming System

INTERVENTIONS:
Device: Bair Paws Patient Adjustable Warming System — Bair Paws system uses forced-air warming. This system will be used for patients randomized to active pre-warming.
  Other Names: Bair Paws Flex Gown

SUMMARY:
The application of active warming to patients whether awake or under general anesthesia has been proven safe in numerous studies and it is common practice to use warmers. The warmers are commonly used with both the supplied blankets and also with hospital blankets.

Subjects receiving standard care will not benefit from this study. Subjects in the investigational group may benefit in several ways:

* Increased comfort in the pre-operative period by being warmer
* Decreased incidence of mild hypothermia
* Possible decreased incidence of transfusion with less bleeding
* Possible decreased pain and discomfort in the Post-Anesthesia Care Unit (PACU)
* Possible shorter stay in the PACU and overall Length of Stay (LOS)
* Possible decreased risk for surgical site infection

ELIGIBILITY:
Inclusion Criteria:

* Elective or "urgent" surgery under general anesthesia
* ≥19 years but ≤85 years of age
* Able to provide informed consent.

Exclusion Criteria:

* Refusal of Informed consent
* Metabolic derangement/drug therapy already affecting thermal homeostasis
* Preexisting hypothermia (<35.5 degreeC) or hyperthermia (>37.5 degreeC) (oral)
* Surgical procedure anticipated to be longer than 6 hours or less than 1 hour
* Emergency (category 1a) Surgery
* Patients undergoing exclusively spinal or epidural anesthesia
* Patients receiving aortic cross-clamping
* Patients receiving transdermal medications

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Duration of hypothermia | Up to 12 hours, until PACU discharge
  The primary endpoint is duration of hypothermia as measured by the area under the curve (AUC). This is achieved by recording patient temperature readings continuously from baseline (prior to initiation of 30 minutes if active or passive pre-warming) until PACU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Merchant, MD, Principal Investigator — Staff Anesthesiologist
Locations (1):
- Royal Columbian Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lau A, Lowlaavar N, Cooke EM, West N, German A, Morse DJ, Gorges M, Merchant RN. Effect of preoperative warming on intraoperative hypothermia: a randomized-controlled trial. Can J Anaesth. 2018 Sep;65(9):1029-1040. doi: 10.1007/s12630-018-1161-8. Epub 2018 Jun 5. PMID 29872966